CLINICAL TRIAL: NCT04590976
Title: Patients' Preferences in the Treatment of Hormone-sensitive Metastatic Prostate Cancer: a Discrete Choice Experiment
Brief Title: Metastatic Prostate Cancer Men's Attitudes Towards Treatment of the Local Tumour and Metastasis Evaluative Research
Acronym: IP5-MATTER
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 276834
Record Dates: First submitted 2020-08-05; First posted 2020-10-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer Metastatic; Radiotherapy Side Effect; Surgery; Urologic Cancer; Quality of Life; Patient Satisfaction; Health Care Utilization
MeSH Terms: conditions — Radiation Injuries; Urologic Neoplasms; Patient Satisfaction; Patient Acceptance of Health Care | interventions — delta 24-sterol reductase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthcare Professionals (n = 5): Intervention: Single, Semi-Structure Interview to identify and define the key attributes associated with treatment options that would warrant trade-off evaluation. These will be used to create the first version of the questionnaire
  Interventions: Other: Semi-Structured Interview Healthcare Professional
- Stage 1 (n = 5): Intervention: Single, Semi-Structure Interview to identify and define the key attributes associated with treatment options that would warrant trade-off evaluation. These will be used to create the first version of the questionnaire
  Interventions: Other: Semi-Structured Interview Patients
- Stage 2 (n = 10): Intervention: Single, "Think Aloud Interview" Interview. These will be analysed using an inductive thematic analysis by at least two researchers. Common themes will be extracted by researchers individually and then discussed and agreed.
  Interventions: Other: Think Aloud Interview Patients
- Stage 3 (n = 300): Intervention: Single, Discrete Choice Experiment Questionnaire at Enrollment Visit
  Interventions: Other: Discrete Choice Experiment (DCE) Patients

INTERVENTIONS:
Other: Semi-Structured Interview Healthcare Professional — Interview
  Groups: Healthcare Professionals (n = 5)
Other: Semi-Structured Interview Patients — Interview
  Groups: Stage 1 (n = 5)
Other: Think Aloud Interview Patients — Interview
  Groups: Stage 2 (n = 10)
Other: Discrete Choice Experiment (DCE) Patients — DCE Questionnaire
  Groups: Stage 3 (n = 300)

SUMMARY:
Systemic therapy (i.e Androgen Deprivation Therapy with Docetaxel, Enzalutamide, Apalutamide or Abiraterone Acetate) has increased overall survival in men with hormone-sensitive metastatic prostate cancer.

Novel local cytoreductive treatments and metastasis directed therapy are being evaluated, these can confer additional harm, but might improve survival.

We aim to elicit men's preferences for and willingness to accept trade-offs between potential improved survival and cytoreductive treatment risks using a 'discrete choice experiment'.

DETAILED DESCRIPTION:
OBJECTIVES: To determine the attributes associated with treatment that are most important to men with hormone-sensitive metastatic prostate cancer (mPCa). To determine men's preferences for, and trade-offs between, the attributes (survival and side-effects) of different treatment options in metastatic prostate cancer including systemic therapy, local and metastases-directed physical therapies.

PHASE: Prospective multi-centre observational cohort

DESIGN: Discrete choice experiment, single-visit, electronic questionnaire design

SAMPLE SIZE: Multi-centre Stage (Stage 3) n = 300 patients

POPULATION: Men with newly-diagnosed metastatic prostate cancer who have not consented to a form of local cytoreductive or metastasis directed therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with prostate cancer within 4 months of screening visit
2. Performance status 0-2

Exclusion Criteria:

1. Castrate-resistant metastatic prostate cancer
2. Patient has consented to a form of local cytoreductive treatment to prostate
3. Patient has consented to a form of metastasis directed therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with newly-diagnosed hormone-sensitive metastatic prostate cancer who have not consented to a form of local cytoreductive or metastasis directed therapy.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Treatment attribute preferences as assessed using a study-specific think aloud interview. | Through study completion, an average of 3 months [Stage 2] (Think Aloud Interview).
  Qualitative work derived from "Think Aloud Interviews". Treatments include radiotherapy, surgery, ablation and metastasis directed therapy.
Willingness to accept treatment attributes, and trade-offs between these, using a study-specific Discrete Choice Experiment (DCE) Questionnaire | Through study completion, an average of 1 year [Stage 3] (Discrete Choice Experiment (DCE) Questionnaire). Trade-off from Marginal Rate of Substitution calculate as percentage points (0 to 100).
  Utility values obtained via multinominal logit estimates from discrete choice experiment

SECONDARY OUTCOMES:
Willingness to accept the potential effect sizes that are shown in trials. | Through study completion, an average of 1 year [Stage 3] (Discrete Choice Experiment (DCE) Questionnaire). No scale.
  Derived from discrete choice experiment finding analysed alongside reported outcomes from ongoing therapeutic trials.

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Ahmed, PhD, FRCS, Principal Investigator — Imperial College London
Locations (35):
- United Kingdom (35):
  - NHS Grampion, Aberdeen
  - Besti Cadwaladr University, Bangor
  - Ysbyty Gwynedd Hospital, Bangor
  - Hamphire Hospitals NHS Foundation Trust, Basingstoke
  - Royal Bath United Hospital, Bath
  - Bedford Hospital, Bedford
  - Royal Bolton Hospital, Bolton
  - Brighton and Sussex hospital, Brighton
  - East Suffolk and North Essex NHS Foundation Trust, Colchester
  - Dartford and Gravsham NHS Trust, Dartford
  - Royal Devon and Exeter Hospital, Exeter
  - Medway NHS Foundation Trust, Gillingham
  - Northern Lincolnshire and Goole NHS Foundation Trust, Grimsby
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - Imperial College London, Hammersmith
  - North Tees and Hartlepool NHS Foundation Trust, Hartlepool
  - West Middlesex University Hospital, Isleworth
  - Queen Elizabeth Hospital, Kings Lynn
  - Kingston Hospital NHS Foundation Trust, Kingston
  - Chelsea and Westminster Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, Chelsea Research Centre, London
  - Luton and Dunstable University Hospital, Luton
  - Wirral University Teaching Hospital Nhs Foundation, Metropolitan Borough of Wirral
  - Freeman Hospital, Newcastle, Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospital, Nottingham
  - University Hospitals Dorset NHS Foundation Trust, Poole
  - East Surrey Hospital, Redhill
  - Royal Shrewsbury Hospital, Shrewsbury
  - Southampton General Hospital, University Hospital Southampton NHS Foundation Trust (UHS), Southampton
  - East and North Hertfordshire Nhs Trust, Stevenage
  - Sunderland Royal Hospital, City Hospitals Sunderland NHS Foundation Trust, Sunderland
  - Musgrove Park Hospital - Somerset NHS Foundation Trust, Taunton
  - The Royal Cornwall Hospital, Truro
  - Wrexham Maelor, Wrexham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Connor MJ, Genie MG, Gonzalez M, Sarwar N, Thippu Jayaprakash K, Horan G, Hosking-Jervis F, Klimowska-Nassar N, Sukumar J, Pokrovska T, Basak D, Robinson A, Beresford M, Rai B, Mangar S, Khoo V, Dudderidge T, Falconer A, Winkler M, Watson V, Ahmed HU. Metastatic prostate cancer men's attitudes towards treatment of the local tumour and metastasis evaluative research (IP5-MATTER): protocol for a prospective, multicentre discrete choice experiment study. BMJ Open. 2021 Nov 18;11(11):e048996. doi: 10.1136/bmjopen-2021-048996. PMID 34794989